CLINICAL TRIAL: NCT06937138
Title: Comparison of AI-Assisted vs Surgeon-Planned Trajectories in Freehand Femoral Neck Screw Fixation: A Multicenter Randomized Controlled Trial
Brief Title: Artificial Intelligence-Assisted vs Surgeon-Planned Trajectories in Freehand Femoral Neck Screw Fixation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Fawwaz Al-Smadi, MD, Medical doctorate student, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025.0198-01
Record Dates: First submitted 2025-04-18; First posted 2025-04-22 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Femoral Neck Fractures
Keywords: Screw Placement Accuracy; Artificial Intelligence in Surgical Planning; Femoral Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, prospective, randomized controlled trial (RCT) designed to evaluate the effectiveness and safety of artificial intelligence (AI)-assisted versus surgeon-directed screw trajectory planning in freehand percutaneous internal fixation of femoral neck fractures. To obtain 266 evaluable patients, a total of 334 participants will be enrolled, accounting for an anticipated 20% dropout rate. Eligible patients will be randomly assigned in a 1:1 ratio to either the AI-assisted screw path planning group (n = 167) or the surgeon-directed screw path planning group (n = 167).
  All patients in both groups will undergo the same standardized freehand cannulated screw fixation procedure and will receive uniform perioperative care, rehabilitation guidance, and scheduled follow-up assessments throughout the 12-month study period.
Who Masked: Participant, Outcomes Assessor
Masking Description: In addition to outcome assessors, third-party orthopedic specialists responsible for postoperative evaluation of screw trajectory accuracy will also be masked to group allocation. These blinded experts will independently assess the appropriateness and accuracy of screw placement in cases where discrepancies arise between AI-recommended and surgeon-modified trajectories. This masking ensures objective evaluation and minimizes assessment bias in the radiographic analysis of screw positioning.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI-Assisted Screw Path Planning Group (Experimental): In the AI-assisted group, the trajectory for screw placement during femoral neck fracture fixation will be guided by an AI algorithm based on intraoperative X-ray imaging. The system will automatically suggest the screw entry point and trajectory, which are displayed for the surgeon to follow during freehand guidewire insertion under fluoroscopy. The surgeon will proceed with the operation after confirming the feasibility of the AI-generated plan. In principle, surgeons are advised not to modify the AI-recommended trajectory unless necessary, to preserve the independent evaluative value of the AI-assisted plan. If significant disagreement arises between the surgeon's judgment and the AI-recommended trajectory, a third-party orthopedic specialist-blinded to group allocation-will conduct an independent postoperative assessment of the screw placement's appropriateness and accuracy.
  Interventions: Procedure: AI-Assisted Screw Path Planning
- Surgeon-Directed Screw Path Planning Group (Active Comparator): In the surgeon-directed planning group, the screw trajectory will be determined entirely by the operating surgeon, based on personal experience and interpretation of intraoperative fluoroscopy. All decisions regarding the screw entry point and trajectory will be made manually without assistance from the AI planning module.
  Interventions: Procedure: Surgeon-Directed Screw Path Planning

INTERVENTIONS:
Procedure: AI-Assisted Screw Path Planning — The trajectory for screw placement during femoral neck fracture fixation will be guided by an AI algorithm based on intraoperative X-ray imaging. The system will automatically suggest the screw entry point and trajectory, which are displayed for the surgeon to follow during freehand guidewire insertion under fluoroscopy. The surgeon will proceed with the operation after confirming the feasibility of the AI-generated plan. In principle, surgeons are advised not to modify the AI-recommended trajectory unless necessary, to preserve the independent evaluative value of the AI-assisted plan. If significant disagreement arises between the surgeon's judgment and the AI-recommended trajectory, a third-party orthopedic specialist-blinded to group allocation-will conduct an independent postoperative assessment of the screw placement's appropriateness and accuracy.
  Arms: AI-Assisted Screw Path Planning Group
Procedure: Surgeon-Directed Screw Path Planning — The screw trajectory will be entirely determined manually by the operating surgeon, based on personal experience and interpretation of intraoperative fluoroscopy, without reliance on any AI recommendation module.
  Arms: Surgeon-Directed Screw Path Planning Group

SUMMARY:
The goal of this clinical trial is to compare two different methods of screw path planning-AI-assisted versus surgeon-directed-in freehand percutaneous femoral neck fracture fixation surgery. The study will include adult patients diagnosed with femoral neck fractures who are eligible for cannulated screw fixation under fluoroscopic guidance.The main questions it aims to answer are:

Does AI-assisted screw path planning improve the radiographic accuracy of screw placement (screw deviation, tip position, and inter-screw parallelism)? Does AI-assisted planning reduce operative time, number of intraoperative fluoroscopy exposures, intraoperative blood loss (mL) and surgeon workload compared with surgeon-directed planning? Does AI-assisted planning reduce postoperative complications and improve functional outcomes compared to surgeon-directed planning? Researchers will compare the AI-assisted planning group to the surgeon-directed planning group to determine whether AI guidance contributes to enhanced surgical precision, reduced intraoperative burden, and improved recovery outcomes.

Participants will:

Undergo freehand percutaneous internal fixation of femoral neck fractures with either AI-assisted or surgeon-directed screw path planning, Receive standardized perioperative care and follow-up at defined intervals, Be evaluated through clinical assessments, imaging studies, and documentation of intraoperative and postoperative metrics over a 12-month follow-up period.

DETAILED DESCRIPTION:
Femoral neck fractures, occurring between the femoral head and the base of the femoral neck, are among the most common hip injuries, particularly in the elderly population. While surgical fixation with closed reduction and cannulated screws is a widely accepted standard, challenges such as suboptimal screw placement, prolonged fluoroscopy exposure, and increased risk of complications like nonunion or avascular necrosis persist-largely influenced by surgeon experience and intraoperative variability.

To address these limitations,this trial investigates the effectiveness and safety of artificial intelligence (AI)-assisted versus surgeon-directed screw path planning in freehand percutaneous internal fixation of femoral neck fractures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Radiologically confirmed diagnosis of femoral neck fracture (displaced or non-displaced);
* Scheduled to undergo internal fixation with cannulated screws as the initial treatment strategy during the study period;
* Capable of understanding the study procedures and providing informed consent;
* Willing and able to adhere to the prescribed postoperative follow-up schedule and rehabilitation instructions.

Exclusion Criteria:

* Evidence of avascular necrosis of the femoral head on the affected side prior to surgery;
* Inability to tolerate the surgical intervention;
* Severe physical illnesses, cognitive problems (such as memory loss), or mental health conditions that may impair the ability to comply with medical instructions or attending scheduled follow-up appointments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2025-11-14 (Actual); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-06-15 (Estimated)

PRIMARY OUTCOMES:
Radiographic Accuracy of Screw Placement | Postoperative Day 1
  Accuracy of screw placement assessed on standardized anteroposterior and lateral radiographs.

SECONDARY OUTCOMES:
Number of Fluoroscopy Exposures | Intraoperative
  Total number of C-arm fluoroscopy shots used during screw placement will be recorded and compared between groups.
Operative Time | Intraoperative
  Total surgical time will be recorded and compared between the AI-assisted and surgeon-directed groups.
Intraoperative Blood Loss (mL) | Intraoperative
  Blood loss will be estimated intraoperatively and documented for each case.
Number of Drilling Attempts | Intraoperative
  Total number of drilling attempts required to achieve acceptable guidewire placement.
Surgeon Workload (NASA-TLX) | Immediately after surgery
  Workload evaluated using the NASA Task Load Index, including mental, physical, temporal demand, performance, effort, and frustration subscales.
Functional Recovery - Harris Hip Score (HHS) | 3, 6, and 12 months postoperatively
  Functional outcomes will be evaluated using the Harris Hip Score. Higher scores indicate better function.
Overall complication rate | Up to 12 months
  Composite rate of postoperative complications, including avascular necrosis, nonunion, delayed union, loss of reduction, screw cut-out, hardware failure, need for reoperation, wound complications, and other surgery-related adverse events.

OTHER OUTCOMES:
Surgeon Confidence Score | Immediately after surgery
  Surgeon self-reported confidence in the trajectory planning and screw placement accuracy measured using a 5-point Likert scale.
AI Override / Modification Rate (AI Group Only) | Intraoperative
  Frequency and proportion of cases where the operating surgeon significantly modified or overrode the AI-recommended trajectory, with reasons recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Guohui Liu, MD, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Bobin Mi, MD, PhD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology; Fawwaz Al-Smadi, MD, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (4):
- China (4):
  - Union Hospital, Tongji Medical College, HUST - Jinyinghu International Hospital, Wuhan
  - Union Hospital, Tongji Medical College, HUST - Main Campus, Wuhan
  - Union Hospital, Tongji Medical College, HUST - Orthopedic Hospital, Wuhan
  - Union Hospital, Tongji Medical College, HUST - West Campus, Wuhan

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) underlying the results of this study will be made available upon reasonable request.